CLINICAL TRIAL: NCT00860678
Title: Influence of Regular Physical Activity on Exercise Capacity, Cardiac Remodeling and Endothelial Function in Patients After Aortic Valve Replacement
Brief Title: Physical Activity in Patients After Aortic Valve Replacement (Valve-ex)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Technical University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2152/08
Record Dates: First submitted 2009-03-11; First posted 2009-03-12 (Estimated); Last update posted 2009-03-12 (Estimated); Status verified 2009-03

CONDITIONS: Valvular Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Exercise

ARMS (2):
- A (Active Comparator): Training group
  Interventions: Other: Physical activity
- B (Other): Controls
  Interventions: Other: no Intervention

INTERVENTIONS:
Other: Physical activity
  Arms: A
Other: no Intervention
  Arms: B

SUMMARY:
A structured and supervised, 3-month physical activity intervention in patients after aortic valve replacement due to severe stenosis, accompanied by examination of cardiac size and function, exercise capacity and endothelial function before, three and six months after operation; comparison with a non-intervention control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe valvular aortic stenosis and indication for valve replacement

Exclusion Criteria:

* Coronary heart disease with indication for additional bypass surgery Leading insufficiency of the valve
* Age < 65 or > 75
* Diseases or conditions leading to additional risks during physical activity (e.g. diabetes, arthrosis, obstructive pulmonary disease)

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)

PRIMARY OUTCOMES:
Maximum oxygen uptake

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Prevention and Sports Medicine Technische Universität München, München, Bavaria, Germany

REFERENCES:
- [Derived] Abraham LN, Sibilitz KL, Berg SK, Tang LH, Risom SS, Lindschou J, Taylor RS, Borregaard B, Zwisler AD. Exercise-based cardiac rehabilitation for adults after heart valve surgery. Cochrane Database Syst Rev. 2021 May 7;5(5):CD010876. doi: 10.1002/14651858.CD010876.pub3. PMID 33962483